CLINICAL TRIAL: NCT05934604
Title: Targeting Large-scale Networks in Depression With Real-time fMRI Neurofeedback
Brief Title: Targeting Large-scale Networks in Depression With Real-time fMRI (Functional Magnetic Resonance Imaging) Neurofeedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Stephan F. Taylor, Professor of Psychiatry, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00228741
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants
Keywords: Healthy; fMRI; Neurofeedback

STUDY DESIGN:
Masking Description: Phase 2 is not blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic resonance imaging (MRI) group (Experimental): Healthy volunteers will have two functional magnetic resonance imaging scans (localizer session and the real time functional magnetic resonance imaging neurofeedback session).
  Interventions: Other: Functional magnetic resonance imaging (fMRI)

INTERVENTIONS:
Other: Functional magnetic resonance imaging (fMRI) — Healthy subjects will complete two fMRI sessions after initial assessment and training in the Rest Focus Task (RFT). The first session will be the localizer session to identify the networks involved in switching in the RFT. The second fMRI session, real time functional magnetic resonance imaging neurofeedback (rtfMRI-NF) session, will use localizer information from the first fMRI session to develop a mask for the rtfMRI-NF, and deliver a neurofeedback (NF) stimulus while simultaneously measuring Blood Oxygenation Level Dependent (BOLD) activity for the STOP>RECALL contrast.

SUMMARY:
The purpose of this study is to develop a technique called real time fMRI neurofeedback.

This technique uses a functional MRI scanner, except that special software allows the researchers to measure activity in participants brain, using fMRI, and then give information, in the form of a feedback signal, which indicates brain activity in real time, while in the MRI scanner. The larger goal of this study is to develop ways to help people, including those with depression, better regulate brain activity. The researchers think that this may be helpful in managing psychiatric symptoms.

This study design has three phases, however, only two phases (phase 2 and 3) are considered to be a clinical trial.

Therefore, this registration will include phase 2 at this time.

DETAILED DESCRIPTION:
During the second phase of the project healthy participants (approximately 12) will have three study visits (two fMRIs) over 2-4 weeks.

Note: As the study is a feasibility/development study, alterations of the task design for the primary outcome measures will be done to achieve objectives of developing at task that recruits from the target region (salience network). In phase 1 of the study, changes to the task are ongoing, and the same may occur for phase 2 in order to develop a viable neurofeedback paradigm. Therefore, detailed descriptions of the outcome measures are not entered at this time, as we don't know exactly what those are. When we do, the entry will be updated.

Note: As of 7/26/2024, the study is rolling back from 'Completed' to 'Recruiting' status in order to include more healthy controls and temporarily resume active development of the task design.

ELIGIBILITY:
Inclusion Criteria (phase 2 participants):

* Ability and willingness to give informed consent to participate
* Not taking any medication, prescription or non-prescription, with psychotropic effects (birth control medications allowed)
* If a woman of child-bearing age, not pregnant or trying to become pregnant
* No history of serious neurological illness (including, but not limited to, seizures/epilepsy) or current medical condition that could compromise brain function, such as liver failure
* No history of closed head injury (see protocol for more details)
* Ability to tolerate small, enclosed spaces without anxiety
* No metals, implants or metallic substances within or on the body that might cause adverse effects to the subject in a strong magnetic field, or interfere with image acquisition
* Size compatible with scanner gantry

Exclusion Criteria (phase 2 participants):

- History of past or current mental illness (except for simple phobias), but prior history of substance dependence ok if in remission for greater than 5 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent (BOLD) signal change during the Focus greater (>) Rest contrast during the localizer session | Approximately 40 minutes (during MRI)
BOLD signal change during the Focus>Rest contrast, comparing baseline with transfer runs (no NF in either), during the rtfMRI-NF session | Approximately 40 minutes (during MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Taylor, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No